CLINICAL TRIAL: NCT00715637
Title: Phase III Open-Label Randomized Study of Amonafide L-Malate in Combination With Cytarabine Compared to Daunorubicin in Combination With Cytarabine in Patients With Secondary Acute Myeloid Leukemia (AML)- The ACCEDE Study
Brief Title: Phase III Randomized Study of Amonafide (AS1413) and Cytarabine Versus Daunorubicin and Cytarabine in Patients With Secondary Acute Myeloid Leukemia (AML)- the ACCEDE Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antisoma Research (Industry)
Responsible Party: Bina Tejura/Medical Director, Antisoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 509912; NCT00509912 (obsolete NCT alias)
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Secondary Acute Myeloid Leukemia (Secondary AML, sAML)
Keywords: AML; Leukemia; MDS; Amonafide; Cytarabine; Daunorubicin; Lymphatic disorders
MeSH Terms: conditions — Leukemia; Lymphatic Diseases | interventions — Daunorubicin; Cytarabine; amonafide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Amonafide in Combination with Cytarabine
  Interventions: Drug: Amonafide and Cytarabine
- Arm B (Active Comparator): Daunorubicin in Combination with Cytarabine
  Interventions: Drug: Daunorubicin and Cytarabine

INTERVENTIONS:
Drug: Daunorubicin and Cytarabine — Daunorubicin: 45 mg/m2 over 30 minutes daily on days 1-3 (up to max. of 2 courses) Cytarabine: 200 mg/m2 IV continuous infusion daily on days 1-7 (up to max. of 2 courses)
  Arms: Arm B
Drug: Amonafide and Cytarabine — Amonafide: 600 mg/m2 IV over 4 hours daily on Days 1-5 (up to max. 2 courses) Cytarabine: 200 mg/m2 IV continuous infusion daily on Days 1-7 (up to max. 2 courses)
  Arms: Arm A

SUMMARY:
Amonafide is a DNA intercalating agent and inhibitor of topoisomerase II that has been extensively studied in patients with malignant solid tumors. Amonafide has also been studied in patients with AML.

The purpose of this study is to assess the relative efficacy and safety of amonafide in combination with cytarabine compared to daunorubicin with cytarabine in subjects with documented secondary AML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to WHO diagnostic criteria (at least 20% blasts in the peripheral blood or bone marrow), with FAB classification other than M3 (Acute Promyelocytic Leukemia), documented by bone marrow aspiration and biopsy performed within 14 days prior to administration of 1st dose of remission induction chemotherapy;
* Either: Known and documented exposure to specific leukemogenic therapy of a specified nature for a non-myeloid condition; OR Documented diagnosis of MDS according to WHO criteria for at least 3 months prior to study entry, with prior bone marrow aspirate, biopsy and peripheral blood smear documenting MDS available to be submitted for subsequent central pathology review.
* Age 18 years or older;
* Eastern Cooperative Oncology Group (ECOG) performance score =< 2;
* Fertile sexually active patients (men and women) must use an effective method of contraception which must be continued throughout the study.
* Women of childbearing potential must have a negative serum pregnancy test.
* Left Ventricular Ejection Fraction (LVEF) >= 50%, as determined by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO) within 14 days prior to administration of 1st dose of remission induction chemotherapy;
* Adequate renal function as evidenced by the following laboratory test, obtained within 10 days prior to administration of 1st dose of remission induction chemotherapy: Serum creatinine =< 1.5 x ULN;
* Adequate hepatic function as evidenced by the following laboratory tests, obtained within 10 days prior to administration of 1st dose of remission induction chemotherapy (unless attributed to hepatic involvement with AML): Total serum bilirubin =< 1.5 x ULN;Serum AST and ALT =< 1.5 x ULN;
* Ability of the patient to participate fully in all aspects of this clinical trial;
* Written Informed Consent and HIPAA authorization (USA sites only) must be obtained and documented.

Exclusion Criteria:

* Histologic diagnosis of FAB M3 Acute Promyelocytic Leukemia;
* Clinically active CNS leukemia;
* Prior induction therapy for AML;
* Known HIV positive;
* Known active hepatitis B or C, or any other active liver disease;
* Patients with parenchymal abnormality on screening chest x-ray must have no evidence of pulmonary infection on chest tomography (CT) prior to starting remission induction therapy.
* Any major surgery or radiation therapy within 4 weeks prior to study entry;
* Prior cytotoxic chemotherapy for MDS within 4 weeks prior to study entry (patients with rapidly rising blast count may be enrolled within 4 weeks of prior cytotoxic chemotherapy with waiver from the Medical Monitor);
* Persistent chronic non-hematologic toxicity (other than alopecia) greater than grade 1 from prior therapy for MDS;
* Serious concomitant illnesses (for example, pulmonary infiltrate, unstable angina or myocardial infarction or stroke within 3 months prior to study entry, congestive heart failure AHA class 2 or greater, uncontrolled hypertension, uncontrolled diabetes, actively bleeding gastric ulcer, etc.), which in the investigator's opinion would not make the patient a good candidate for the trial;
* Pregnant or breast feeding;
* History of clinically significant allergic reactions attributed to compounds of similar chemical or biological composition to amonafide, cytarabine or daunorubicin;
* Prior enrollment in this trial;
* Any other known condition (e.g., familial, sociological, or geographical) or behavior (including substance dependence or abuse, psychological or psychiatric illness), which in the investigator's opinion would make the patient a poor candidate for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Rate of CR + CRi (which includes CRc and CRd) will be determined by assessing the proportion of patients who achieved CR or CRi among all evaluable patients. | Course 1/Course 2 Day 37 bone marrow assessments and confirmation bone marrow 30 days later

SECONDARY OUTCOMES:
Median duration of remission and median duration of disease free survival. | Follow-up visits following post-remission therapy

CONTACTS AND LOCATIONS:
Locations (158):
- United States (30):
  - UCLA Medical Center, Los Angelas, California
  - Univ of Southern California Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - The Blood and Marrow Transplant Group of GA, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals, Iowa City, Iowa
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - LSU Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Michigan State University, Lansing, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northshore Hospital - Monter Cancer Center, Lake Success, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Taussig Cancer Center, Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Intermountain Healthcare, Salt Lake City, Utah
- Argentina (5):
  - Hospital Italiano de La Plata, Buenos Aires
  - Hospital General de Agudos "Dr. Teodoro Alvarez", Ciudad Autónoma de Bs. As.
  - Clinical Hematology Service, Ciudad Autónoma de Bs. As.
  - Hospital Provincial de Cordoba, Córdoba
  - Sanatorio Parque, Rosario - Santa Fe
- Australia (8):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (3):
  - LKH-Universitats Klinikum Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
  - Landesklinikum St. Polten, Sankt Pölten
- Belgium (4):
  - University Hospital Gent, Ghent, Gent
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - UCL de Mont-Godinne, Yvoir
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - QEII Center for Clinical Research, Halifax
  - The Ottawa Hospital - General Campus, Ottawa
- Chile (3):
  - Hospital Santa Maria, Santiago
  - Hospital DIPRECA, Santiago
  - Hospital Dr. Gustavo Fricke, Viña del Mar
- Czechia (3):
  - University Hospital Kralovske Vinohrady Prague, Prague
  - General University Hospital Prague, Prague
  - Institute of Haematology and Blood Transfusion Prague, Prague
- Ecuador (3):
  - Instituto Ecuatoriano de Seguridad Social Hospital Regional Teodoro Maldonado Carbó, Guayaquil
  - Hospital Carlos Andrade Marin, Quito
  - Hospital Militar, Quito
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (6):
  - Hopital de Versailles, Versailles, Le Cheaney
  - Hopital Sud, Amiens
  - Hopital Edouard Herriot, Lyon
  - Hopital-DIEU, Paris
  - Hopital du Haut Leveque, Pessac
  - Hopital Bretonneau - CHRU de Tours, Tours
- Germany (12):
  - Charite - Campus Benjamin Franklin, Berlin
  - Campus Virchow Klinikum, Berlin
  - Evangelische Kliniken GmbH, Bonn
  - St Antonius Hospital, Eschweiler
  - Universitatsklinikum Essen, Essen
  - Stadtische Kliniken Frankfurt, Frankfurt
  - Asklepios Kliniken Altona, Hamburg
  - Medizin Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum Leverkusen, Leverkusen
  - Markische Kliniken GmbH Klinikim Ludenscheid, Lüdenscheid
  - Universitätsmedizin Mannheim, Mannheim
- Hungary (4):
  - Szent Istvan and Szent Laszlo Corporate Hospital - Out-patient Clinic of the Municipality Government, Budapest
  - Petz Aladar County Teaching Hospital, Győr
  - Kaposi Mór County Teaching Hospital, Kaposvár
  - University of Pecs, Pécs
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - University of Brescia, Brescia
  - A.O.U Careggi, Florence
  - A.O.U San Martino, Genova
  - A.O. Cardarelli, Napoli
  - A.O. San Salvatore, Pesaro
  - A.O.U Pisana Santa Chiara, Pisa
  - Università degli Studi di Roma "La Sapienza", Roma
  - Ospedale S. Eugenio, Rome
  - Istituto Clinico Humanitas, Rozzano
- Poland (9):
  - Teaching Hospital of the Medical University in Bialystok, Bialystok
  - Academic Clinical Centre - Teaching Hospital of the Medical University of Gdansk, Gdansk
  - Nicolaus Copernicus Provincial Specialist Hospital in Lodz, Lodz
  - Provincial Hospital in Opole, Opole
  - Poznan Stare Miasto Health Care Facility, Poznan
  - Janusz Korczak Provincial Specialist Hospital, Słupsk
  - Military Institue of Health Services, Warsaw
  - Institute of Hematology and Transfusiology, Warsaw
  - Independent Public University Hospital No. 1 in Wroclaw, Wroclaw
- Romania (6):
  - Dr. Constantin Opris County Emergency Hospital, Internal Medicine Department, Baia Mare
  - Brasov County Emergency Clinical Hospital, Brasov
  - Colentina Clinical Hospital, Internal Medicine Department, Bucharest
  - Fundeni Clinical Institute "Stefan Berceanu" Center for Hematology and Bone Marrow Transplant, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - Sibiu County Clinical Hospital, Internal Clinic II, Sibiu
- Russia (13):
  - State Medical Institution Republican Hospital n.a. V.A. Baranov, Petrozavodsk, Republic of Karelia
  - Municipal Medical Institution Municipal Hospital #1, Cherepovets
  - State Medical Institution Irkutsk Regional Clinical Hospital, Irkutsk
  - State Medical Institution Territorial Clinical Hospital #1, Khabarovsk
  - State Medical Institution Territorial Clinical Oncological Center, Krasnodar
  - State Institution Russian Oncological Research Center n.a. N.N. Blokhin of the Russian Academy of Medical Sciences, Moscow
  - Moscow State Medical Institution Municipal, Moscow
  - Municipal Medical Institution, Perm
  - State Higher Educational Instution Rostov State, Rostov-on-Don
  - State Medical Institution Leningrad Regional Clinical Hospital, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University n.a. I.P. Pavlov under the Federal Agency for Healthcare and Social Development, Saint Petersburg
  - Federal Center of Heart, Blood and Endocrinology, Saint Petersburg
  - State Medical Institution Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- South Korea (7):
  - Inje University Busan Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital in YUHS, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic I Provinicial, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario La Fe, Valencia
- Taiwan (7):
  - Chang Gung Memorial Hospital Kao Hsiung Branch, Niao-Sung Hsiang, Kaohsiung Hsien
  - Changhua Christian Hospital (CCH), Changhua
  - Chinese Medical University Hospital (CMUH), Taichung
  - National Cheng Kung University Hospital (NCKUH), Tainan
  - National Taiwan University Hospital (NTUH), Taipei
  - Mackay Memorial Hospital, Taipei
  - Veterans General Hospital Taipei (VGH-TP), Taipei
- Ukraine (10):
  - Public Institution 'Cherkasy Regional Oncology Center', Cherkasy
  - Dnipropetrovsk City General Clinical Hospital #4, Dnipropetrovsk
  - Ivano-Frankivsk State Medical University, Ivano-Frankivsk
  - Khmelnytsky Regional Hospital, Khmelnytsky
  - State Institution 'Institute of Blood Pathology and Transfusion Medicine under the UAMS', Lviv
  - Mykolaiv Regional Clinical Hospital, Mykolaiv
  - Odesa Regional Clinical Hospital, Odesa
  - Ukrainian Medical Academy of Dentistry, Poltava
  - M.I. Pyrohov Vinnytsya Regional Clinical Hospital, Vinnytsia
  - O.F. Herbachevsky Zhytomyr Regional Clinical Hospital, Zhytomyr
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, Wales
  - King's College Hospital, London
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Stone RM, Mazzola E, Neuberg D, Allen SL, Pigneux A, Stuart RK, Wetzler M, Rizzieri D, Erba HP, Damon L, Jang JH, Tallman MS, Warzocha K, Masszi T, Sekeres MA, Egyed M, Horst HA, Selleslag D, Solomon SR, Venugopal P, Lundberg AS, Powell B. Phase III open-label randomized study of cytarabine in combination with amonafide L-malate or daunorubicin as induction therapy for patients with secondary acute myeloid leukemia. J Clin Oncol. 2015 Apr 10;33(11):1252-7. doi: 10.1200/JCO.2014.57.0952. Epub 2015 Mar 2. PMID 25732165
- [Derived] Lindsley RC, Mar BG, Mazzola E, Grauman PV, Shareef S, Allen SL, Pigneux A, Wetzler M, Stuart RK, Erba HP, Damon LE, Powell BL, Lindeman N, Steensma DP, Wadleigh M, DeAngelo DJ, Neuberg D, Stone RM, Ebert BL. Acute myeloid leukemia ontogeny is defined by distinct somatic mutations. Blood. 2015 Feb 26;125(9):1367-76. doi: 10.1182/blood-2014-11-610543. Epub 2014 Dec 30. PMID 25550361